CLINICAL TRIAL: NCT00110032
Title: Microenvironment: Imaging/Implications in Brain Tumors; A Preliminary Investigation of the Biodistribution of [F-18]-EF5 in Patients With Brain Tumors
Brief Title: Positron Emission Tomography Using Fluorine F 18 EF5 to Find Oxygen in Tumor Cells of Patients Who Are Undergoing Surgery or Biopsy for Newly Diagnosed Brain Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2012-02651; UPCC 01304; CDR0000423313 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Central Nervous System Germ Cell Tumor; Adult Choroid Plexus Tumor; Adult Craniopharyngioma; Adult Diffuse Astrocytoma; Adult Ependymoblastoma; Adult Ependymoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Grade I Meningioma; Adult Grade II Meningioma; Adult Grade III Meningioma; Adult Medulloblastoma; Adult Meningeal Hemangiopericytoma; Adult Mixed Glioma; Adult Myxopapillary Ependymoma; Adult Oligodendroglioma; Adult Pilocytic Astrocytoma; Adult Pineoblastoma; Adult Pineocytoma; Adult Subependymoma; Adult Supratentorial Primitive Neuroectodermal Tumor (PNET); Meningeal Melanocytoma
MeSH Terms: conditions — Astrocytoma; Ependymoma; Oligodendroglioma; Choroid Plexus Neoplasms; Craniopharyngioma; Neuroectodermal Tumors, Primitive; Glioblastoma; Gliosarcoma; Meningioma; Medulloblastoma; Glioma; Pinealoma; Glioma, Subependymal | interventions — Surgical Procedures, Operative; Congresses as Topic; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

ARMS (3):
- Group 1 (fluorine F 18 EF5, PET) (Experimental): Patients receive fluorine F 18 EF5 (^18F-EF5) IV followed by whole brain and whole body PET scanning OR whole body PET scanning only. Patients then receive nonradioactive EF5 IV over 1-2 ½ hours.
  Interventions: Procedure: conventional surgery; Procedure: positron emission tomography; Radiation: fluorine F 18 EF5; Other: pharmacological study
- Group 2 (EF5, PET) (Experimental): Patients receive nonradioactive EF5 IV over 1-2½ hours followed by ^18F-EF5 IV. Patients then undergo whole brain and whole body PET scanning.
  Interventions: Drug: EF5; Procedure: conventional surgery; Procedure: positron emission tomography; Other: pharmacological study
- Group 3 (EF5, PET) (Experimental): Patients receive nonradioactive EF5 and ^18F-EF5 as in group 2. Patients then undergo whole brain PET scanning.
  Interventions: Drug: EF5; Procedure: conventional surgery; Procedure: positron emission tomography; Radiation: fluorine F 18 EF5; Other: pharmacological study

INTERVENTIONS:
Drug: EF5 — Given IV
  Arms: Group 2 (EF5, PET); Group 3 (EF5, PET)
Procedure: conventional surgery — Undergo surgery
  Other Names: surgery, conventional
Procedure: positron emission tomography — Undergo PET
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Radiation: fluorine F 18 EF5 — Given IV
  Other Names: 18F-EF5
  Arms: Group 1 (fluorine F 18 EF5, PET); Group 3 (EF5, PET)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects of fluorine F18 EF5 when given during positron emission tomography to find oxygen in tumor cells of patients who are undergoing surgery or biopsy for newly diagnosed brain tumors. Diagnostic procedures using fluorine F 18 EF5 and positron emission tomography to detect tumor hypoxia may help in planning cancer treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety of fluorine F 18 EF5 (^18F-EF5) in patients with newly diagnosed brain tumors undergoing surgery or biopsy.

Secondary I. Determine the pharmacokinetics and biodistribution of ^18F-EF5 administered before and after nonradioactive EF5 in these patients.

II. Determine the ability of positron emission tomography (PET) scanning using ^18F-EF5 to detect tumor hypoxia in these patients.

III. Determine the presence and pattern of nonradioactive EF5 binding by immunohistochemistry (IHC) and/or flow cytometry in these patients.

IV. Correlate tumor hypoxia, as measured by PET scanning using ^18F-EF5, with EF5 staining by IHC and/or flow cytometry and recurrence-free survival of these patients.

OUTLINE: Patients are assigned to 1 of 3 groups.

Group 1: Patients receive fluorine F 18 EF5 (^18F-EF5) IV followed by whole brain and whole body positron emission tomography (PET) scanning OR whole body PET scanning only. Patients then receive nonradioactive EF5 IV over 1-2 ½ hours.

Group 2: Patients receive nonradioactive EF5 IV over 1-2½ hours followed by ^18F-EF5 IV. Patients then undergo whole brain and whole body PET scanning.

Group 3: Patients receive nonradioactive EF5 and ^18F-EF5 as in group 2. Patients then undergo whole brain PET scanning. Approximately one day after EF5 administration, all patients undergo surgery or biopsy of the tumor AND biopsy of normal skin adjacent to the incision.

Patients are followed at 2-4 weeks and 4-6 weeks after EF5 administration and then every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and/or clinical and imaging evidence of a de novo mass that is likely to be a brain tumor
* Amenable to debulking surgery or surgical resection or biopsy as standard initial therapy for the tumor
* Performance status - Karnofsky 70-100%
* At least 3 months
* WBC count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin < 1.2 mg/dL
* Creatinine < 1.3 mg/dL
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No other significant cardiac condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study participation
* Weight ≤ 130 kg
* No peripheral neuropathy ≥ grade 3
* No history of allergic reaction attributed to metronidazole
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No other medical condition that would preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-06; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Safety of F-18-EF5 based on the NCI CTCAE version 3.0 | Up to 3 years
  Summarized in descriptive statistics.

SECONDARY OUTCOMES:
Pharmacokinetics of radioactively labeled [F-18]-EF5 | Day 1
Extent of hypoxia, determined by [F-18]-EF5 PET imaging | Up to day 1
IHC analysis of cold EF5 | Up to day 1
Progression-free survival | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Michael Hahn, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States